CLINICAL TRIAL: NCT07240025
Title: Anatomical Determinants and Outcomes of Small Annulus Patients Undergoing TAVR in Different ASIAN Ethnicity
Status: Enrolling by invitation | Type: Observational
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Collaborators: Sarawak Heart Centre (Other); King Chulalongkorn Memorial Hospital (Other); Ramathibodi Hospital (Other); University Malaysia Sarawak (Other); St. Luke's Medical Center, Philippines (Other); Sapporo Heart Center (Unknown)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Clinical Assistant Professor, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: ADAPT-ASIAN
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- AS TAVI patient in Prince of Wales Hospital
- AS TAVI patient in Sarawak Heart Centre/University Malaysia Sarawak
- AS TAVI patient in National Heart Centre Malaysia
- AS TAVI patient in King Chulalongkorn Memorial Hospital
- AS TAVI patient in Ramathibodi Hospital
- AS TAVI patient in St. Luke's Medical Cente
- AS TAVI patient in Sapporo Cardiovascular Clinic

SUMMARY:
Transcatheter aortic valve implantation (TAVI) presents unique challenges for Asian patients compared to Caucasians, largely due to the prevalence of small aortic annulus (SAA) defined based on Caucasians' data (430 mm²), bicuspid aortic valve (BAV), and substantial calcium deposits. No universally accepted cutoff value for defining SAA exists among Asian patients, who tend to have smaller body-built, resulting in inconsistencies across various studies. For the new-generation 20-/23-mm balloon expandable valve, a SAA is categorized as <330 mm². Additionally, Asian Japanese patients have been identified to have extremely SAA (<314 mm²), associated with unexpectedly larger residual transvalvular gradients following TAVI.

Previous research on patient prosthesis mismatch (PPM) impact within the Asian population has also shown inconsistency. The OCEAN-TAVI registry with 1,546 Japanese patients found no significant differences in one-year all-cause and cardiovascular mortality between PPM and non-PPM groups. A study on the Sapien 3 balloon expandable valve in patients with SAA (<430 mm²) found comparable clinical outcomes to non-SAA patients up to five years post-procedure, consistent with findings from a South Korean study. However, a Taiwan study involving 201 patients with PPM indicated higher rates of adverse outcomes at mid-term follow-up. Moreover, TAVI with self-expanding valves (SEV) has shown improved hemodynamic outcomes and reduced PPM incidence compared to balloon expandable valves (BEV) in patients with extreme SAA.

To date, research on inter-racial differences in TAVI among Asian populations is lacking. This multicenter registry aims to evaluate SEV versus BEV outcomes in diverse Asian patients, particularly those with extreme SAA, and to address ethnic-specific challenges in TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Aortic Stenosis patients treated with Transcatherter Aortic Valve Intervention

Exclusion Criteria:

* Transcatherter Aortic Valve Intervention for pure Aortic Regurgitation
* Emergent procedure for any reason;
* Previous aortic valve replacement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective data collection will be carried out at multiple TAVI sites in Asia. Patients with severe AS who underwent TAVI (SEV/ BEV) will be identified from retrospective records (Physical/ Electronic). Consecutive patients who underwent pre-procedural computed tomography (CT) scans for aortic valve evaluation from 2018-1-1 to 2024-12-31 were included.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Bioprosthetic Structural Valve Dysfunction (SVD) at 12 months | 12 months Post-Operation

SECONDARY OUTCOMES:
Mortality rate | Mortality of patients 12 months post-operation
Disabling stroke rate | Rate of disabling stroke 12 months post-operation
Heart failure re-hospitalization rate | Heart failure re-hospitalization rate at 12 month post-operation
Rate of moderate prosthesis-patient mismatch (PPM) | Rate of moderate prosthesis-patient mismatch (PPM) at 12 month post-operation
  In patients with a body mass index <30 kg/m2, PPM was defined as none or mild if the indexed EOA (iEOA) was>0.85 cm2/m2, moderate if the iEOA was 0.85-0.66 cm2/m2 and severe if the iEOA was ≤0.65 cm2/m2. In patients with a body mass index ≥30 kg/m2, PPM was defined as none or mild if the iEOA was>0.70 cm2/m2, moderate if the iEOA was 0.56-0.70 cm2/m2 and severe if the iEOA was ≤0.55 cm2/m2
Rate of severe prosthesis-patient mismatch (PPM) | Rate of severe prosthesis-patient mismatch (PPM) at 12 month post-operation
Device success rate | Device success rate at 30-days post-operation
Device safety rate | Device safety rate at 30-days post-operation
Rate of Bioprosthetic Structural Valve Dysfunction | Bioprosthetic Structural Valve Dysfunction (SVD) at follow-up
Rate of endocarditis | Rate of endocarditis at 12 month
Rate of Non-structural valve dysfunction (NSVD) | Rate of Non-structural valve dysfunction (NSVD) at 12 month
  ≥Moderate aortic regurgitation rate of moderate or severe PPM (PPM: In patients with a body mass index <30 kg/m2, PPM was defined as none or mild if the indexed EOA (iEOA) was>0.85 cm2/m2, moderate if the iEOA was 0.85-0.66 cm2/m2 and severe if the iEOA was ≤0.65 cm2/m2. In patients with a body mass index ≥30 kg/m2, PPM was defined as none or mild if the iEOA was>0.70 cm2/m2, moderate if the iEOA was 0.56-0.70 cm2/m2 and severe if the iEOA was ≤0.55 cm2/m2, PVL, and DVI (severe <0.25, moderate 0.25-0.5, mild >0.5)

CONTACTS AND LOCATIONS:
Overall Officials: Chak Yu Kent So, Clinicnal Assistant Professor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided